CLINICAL TRIAL: NCT06681064
Title: Breast Cancer Evolution During Neoadjuvant Systemic Therapy
Acronym: BELIEVE
Status: Recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5868
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer; ER+ Breast Cancer; HER2+ Breast Cancer
Keywords: Neoadjuvant Therapy
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples Blood samples Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BELIEVE is a translational research study that aims to collect samples of breast cancer tissue and blood from individuals undergoing breast cancer treatment (such as chemotherapy, targeted therapy and immunotherapy) before surgery. In certain cases, MRI scans and stool samples will also be obtained before and during treatment. The samples collected from this study will be used for molecular and genetic research to understand why some cancers respond very well to anticancer treatments, and some do not, develop novel ways of accurately measuring response during treatment, as well as identify which patients are at a higher risk of the cancer coming back after surgery.

DETAILED DESCRIPTION:
Breast cancer is the most common female cancer in the UK and remains one of the leading causes of cancer death. Survival rates have greatly improved over the past forty years due to improvements in early diagnosis, surgical techniques, effective chemotherapy treatments, hormonal therapy, and the introduction of targeted biological treatments. However, despite this, breast cancer continues to be the 4th most common cause of cancer death in the UK and 20% of women diagnosed with this disease do not survive more than ten years after diagnosis.

Systemic anticancer treatments (that is, oral or intravenous treatments such as chemotherapy, targeted therapy and immunotherapy) are routinely given before surgery (called neoadjuvant therapy) in patients with aggressive early and locally advanced breast cancer in order to shrink the cancer and make it more operable. As a result, women receiving neoadjuvant therapy often require less radical surgery to remove their cancer. Clinical trials have shown that the timing of systemic therapy (that is, whether it is given before or after surgery), does not make a difference to survival, and because of this systemic therapy before surgery is now a mainstay of breast cancer treatment.

Clinical trials have also shown that the level of response in both primary breast tumour and nearby lymph nodes to systemic anticancer therapy are strongly associated with cancer relapse and survival. The presence of extensive cancer at the time of surgery is associated with a higher risk of metastatic relapse and a poor prognosis.

This study will deeply analyse samples from a patient's tumour, blood, and stool, as well as data from MRI images, to identify specific features of either the patient or their cancer which could be used to predict whether (a) a treatment is likely to work and (b) once started, whether the treatment is still working. All this data will be combined together to build predictors that can identify: (a) patients who are not responding to therapy and could be directed towards different treatments and (b) patients who are responding very well to treatment and might benefit from therapy de-escalation.

Additionally, by profiling these breast cancers in great detail, this project will allow us to identify new cancer vulnerabilities and drug targets that could then be used for treatment in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-metastatic invasive breast cancer.
2. Be suitable for, but have not commenced, neoadjuvant chemotherapy, targeted therapy, or immunotherapy.
3. If HER2-, suitable for treatment with upfront taxane chemotherapy. If HER2+, suitable for treatment with anti-HER2 targeted therapy.
4. Be aged 18 years and over.
5. Have given written informed consent to participate.

Exclusion Criteria:

1. Metastatic breast cancer at diagnosis.
2. Treatment with neoadjuvant endocrine therapy only.
3. Presence of any psychological, familial or sociological condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early breast cancer patients suitable for neoadjuvant chemotherapy, targeted therapy, or immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2034-05 (Estimated); Study Completion 2034-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients recruited undertaking sequential tumour biopsies, blood samples, and MRI. | Total 10 year recruitment period
Proportion of patients undergoing study procedures within time frames specified by protocol. | Total 10 year recruitment period

SECONDARY OUTCOMES:
Characterisation of serial molecular and imaging tumour and host profiles and correlation with clinical characteristics, treatment responses and patient outcomes. | Total 10 year recruitment period
Integration of multiplatform profiling data to develop predictors of response to therapy. | Total 10 year recruitment period

CONTACTS AND LOCATIONS:
Overall Officials: Stephen-John Sammut, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Background] Sammut SJ, Crispin-Ortuzar M, Chin SF, Provenzano E, Bardwell HA, Ma W, Cope W, Dariush A, Dawson SJ, Abraham JE, Dunn J, Hiller L, Thomas J, Cameron DA, Bartlett JMS, Hayward L, Pharoah PD, Markowetz F, Rueda OM, Earl HM, Caldas C. Multi-omic machine learning predictor of breast cancer therapy response. Nature. 2022 Jan;601(7894):623-629. doi: 10.1038/s41586-021-04278-5. Epub 2021 Dec 7. PMID 34875674